CLINICAL TRIAL: NCT00565461
Title: A Phase 2, Randomized, Open-Label Study to Compare the Immunogenicity and Safety of a Self-Administered LT Vaccine Patch With an LT Vaccine Patch Administered by a Clinician
Brief Title: LT Vaccine Patch Self-Administration Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intercell USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ELT203
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Prevention of Travelers' Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): 40 subjects will have skin prepared using SPS:Buffer and will receive 37.5ug LT patch on the left deltoid by a Clinician on Day 0. Two weeks later will have the same treatment repeated on the right deltoid by the clinician
  Interventions: Biological: heat-labile enterotoxin of E. coli (LT)
- Group 2 (Experimental): 40 subjects will be pretreated with SPS:Buffer and a patch containing 37.5ug will be applied on the left deltoid by the Clinician. Fourteen days later, the same procedure will occur on the left thigh by the clinician.
  Interventions: Biological: heat-labile enterotoxin of E. coli (LT)
- Group 3 (Experimental): 40 subjects will have skin prepared using SPS:Buffer and will receive 37.5ug LT on the left deltoid by the clinician. Two weeks later subject will have the same treatment repeated by self-application in the clinic on the left thigh.
  Interventions: Biological: heat-labile enterotoxin of E. coli (LT)
- Group 4 (Experimental): 40 subjects will have skin prepared using SPS:Buffer and will have 37.5ug LT patch on the left deltoid by a clinician. Two weeks later subjects will have the same treatment repeated by self-application at home on the left thigh.
  Interventions: Biological: heat-labile enterotoxin of E. coli (LT)

INTERVENTIONS:
Biological: heat-labile enterotoxin of E. coli (LT) — 37.5ug patch applied on either the deltoid or the thigh
  Other Names: TD Vaccine System

SUMMARY:
To evaluate the immune responses achieved following self-administered heat-labile enterotoxin of E. coli (LT) vaccination by transcutaneous immunization compared to the immune responses achieved by clinician-administered vaccination.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible to participate in the study:

* Healthy adult males or females 18-64 years of age with signed Informed Consent.
* Women who are not post-menopausal or surgically sterile must have a negative serum or urine pregnancy test at screening and within 24 hours of each vaccination with understanding (through Informed Consent process) to not become pregnant over the duration of the study, and must agree to employ an effective form of birth control for the duration of the study. Acceptable forms of birth control are: abstinence, hormonal contraceptives (oral, injectable, implant, patch, ring), double-barrier contraceptives (condom or diaphragm, with spermicide), and IUD.

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for participation in the study:

* Laboratory abnormalities [as determined by the Toxicity Grading Scale (grade 1-4)] at laboratory screening
* Abnormalities at physical examination [as determined by the Toxicity Grading Scale (grade 1-4)]
* Known allergies to any component of the vaccine
* Known allergies to adhesives
* Participated in research involving investigational product within 30 days before planned date of first vaccination
* Donated blood or blood products such as plasma within the past 30 days
* Ever received investigational enterotoxigenic E. coli, LT, or LT (R192G) or NasalFlu, Berna Biotech, Ltd
* Ever received cholera toxin or vaccine (e.g. Orochol™, Dukoral™)
* History of traveler's diarrhea in the previous two years
* History of abdominal surgery (excluding C-Section, hysterectomy, cosmetic surgery, liposuction, appendectomy, cholecystectomy, ventral hernia repair, and other surgeries not pertaining to gastrointestinal problems) or history of, or recent acute gastrointestinal (GI) illness
* Positive serology for HIV-1, HIV-2, HBsAg, or HCV
* Medical history of acute or chronic skin disease at vaccination area(s)
* Active skin allergy
* Signs of acute skin infection, sunburn or skin abnormalities at the vaccination area(s) including fungal infections, severe acne, or active contact dermatitis, or a history of keloid formation
* Excessively hirsute at the vaccination area(s) that would interfere with patch adhesion in the opinion of the Investigator
* Visible tattoos or marks (tattoos/scars) at the vaccination area(s) that would prevent appropriate dermatologic monitoring of the vaccination site(s)
* Fever greater than or equal to 38.0°C (100.4°F) at the time of planned vaccination
* Women who are pregnant or breastfeeding
* Acute illness at screening or at baseline; or
* Employee of the investigational site.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Forte, MD, Principal Investigator — Arkansas Medical Research Testing
Locations (3):
- United States (3):
  - Arkansas Medical Research Testing, Little Rock, Arkansas
  - Miami Research Associates, South Miami, Florida
  - Jean Brown Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinician Administered (Deltoid): 40 subjects will have skin prepared using SPS:Buffer and will receive 37.5ug LT patch on the left deltoid by a Clinician on Day 0. Two weeks later will have the same treatment repeated on the right deltoid by the clinician
  heat-labile enterotoxin of E. coli (LT): 37.5ug patch applied on either the deltoid or the thigh
- Clinician Administered (Thigh): 40 subjects will be pretreated with SPS:Buffer and a patch containing 37.5ug will be applied on the left deltoid by the Clinician. Fourteen days later, the same procedure will occur on the left thigh by the clinician.
  heat-labile enterotoxin of E. coli (LT): 37.5ug patch applied on either the deltoid or the thigh
- Self Administered (In-clinic): 40 subjects will have skin prepared using SPS:Buffer and will receive 37.5ug LT on the left deltoid by the clinician. Two weeks later subject will have the same treatment repeated by self-application in the clinic on the left thigh.
  heat-labile enterotoxin of E. coli (LT): 37.5ug patch applied on either the deltoid or the thigh
- Self Administered (Non-clinic): 40 subjects will have skin prepared using SPS:Buffer and will have 37.5ug LT patch on the left deltoid by a clinician. Two weeks later subjects will have the same treatment repeated by self-application at home on the left thigh.
  heat-labile enterotoxin of E. coli (LT): 37.5ug patch applied on either the deltoid or the thigh
Period: Overall Study
Arm/Group | Clinician Administered (Deltoid) | Clinician Administered (Thigh) | Self Administered (In-clinic) | Self Administered (Non-clinic)
Started | 40 | 40 | 40 | 40
Completed | 40 | 39 | 39 | 37
Not Completed | 0 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinician Administered (Deltoid) | Clinician Administered (Thigh) | Self Administered (In-clinic) | Self Administered (Non-clinic) | Total
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (12.21) | 35.0 (11.10) | 38.1 (11.18) | 34.1 (11.18) | 36.0 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 21 | 27 | 23 | 99
  Male | 12 | 19 | 13 | 17 | 61
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 40 | 40 | 160

OUTCOME MEASURES:

1. Primary Outcome: GMTs After a Self-administered LT Vaccine Patch (In-clinic or Away From Clinic) Compared to a Clinician-administered LT Vaccine Patch.
Description: The primary endpoint of this trial was to compare the immunogenicity (i.e., GMTs, GMFRs and seroconversion rates for LT IgG and IgA) of subject self-administered [second] vaccination with clinician-administered [second] vaccination, using the deltoid/thigh (Vaccination 1/Vaccination 2) treatment regimen.
  GMT: geometric mean titer
Time Frame: Day 0, Day 14, Day 21, Day 28, Day 35, Day 194
Population: intent to treat population = primary analysis population; defined as all study subjects who were consented, randomized, and had a baseline serology
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titers
Groups:
- Clinician Administered (Deltoid/ Thigh): 1. st vaccination: administered by clinician; location: deltoid
  2. nd vaccination: administered by clinician; location: thigh
- Self Administered (In-clinic & Non-clinic): 1. st vaccination: administered by clinician; location: deltoid
  2. nd vaccination: self-administration either in-clinic or away from the clinic; location: thigh
Arm/Group | Clinician Administered (Deltoid/ Thigh) | Self Administered (In-clinic & Non-clinic)
Number analyzed (Participants) | 41 | 80
geometric mean titers
  LT IgG GMTs - Day 0 | 362 [264 to 496] | 442 [354 to 552]
  LT IgG GMTs - Day 14 | 1974 [1196 to 3258] | 2896 [2032 to 4127]
  LT IgG GMTs - Day 21 | 4747 [3232 to 6973] | 7545 [5759 to 9886]
  LT IgG GMTs - Day 28 | 11153 [8255 to 15068] | 12180 [9832 to 15089]
  LT IgG GMTs - Day 35 | 12165 [9320 to 15877] | 12745 [10519 to 15442]
  LT IgG GMTs - Day 194 | 4997 [3753 to 6654] | 6035 [4917 to 7409]
  LT IgA GMTs - Day 0 | 54 [41 to 69] | 53 [44 to 64]
  LT IgA GMTs - Day 14 | 218 [142 to 335] | 365 [270 to 494]
  LT IgA GMTs - Day 21 | 430 [309 to 598] | 639 [507 to 806]
  LT IgA GMTs - Day 28 | 632 [462 to 864] | 768 [615 to 960]
  LT IgA GMTs - Day 35 | 548 [397 to 757] | 712 [564 to 898]
  LT IgA GMTs - Day 194 | 254 [190 to 341] | 287 [233 to 354]

2. Primary Outcome: GMFR After a Self-administered LT Vaccine Patch (In-clinic or Away From Clinic) Compared to a Clinician-administered LT Vaccine Patch.
Description: The primary endpoint of this trial was to compare the immunogenicity (i.e., GMTs, GMFRs and seroconversion rates for LT IgG and IgA) of subject self-administered [second] vaccination with clinician-administered [second] vaccination, using the deltoid/thigh (Vaccination 1/Vaccination 2) treatment regimen.
  GMFR: geometric mean fold ratio GMFRs relative to the baseline titer were determined for LT IgG and LT IgA at each post-baseline time point. All GMFRs were based on log10-transformed data.
Time Frame: Day 14, Day 21, Day 28, Day 35, Day 194
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: geometric mean fold ratio
Arm/Group | Clinician Administered (Deltoid/ Thigh) | Self Administered (In-clinic & Non-clinic)
Number analyzed (Participants) | 41 | 80
geometric mean fold ratio
  LT IgG GMFR - Day 14 | 6 [4 to 8] | 7 [5 to 9]
  LT IgG GMFR - Day 21 | 14 [9 to 20] | 17 [13 to 23]
  LT IgG GMFR - Day 28 | 31 [22 to 44] | 28 [21 to 36]
  LT IgG GMFR - Day 35 | 34 [23 to 49] | 29 [22 to 38]
  LT IgG GMFR - Day 194 | 14 [10 to 20] | 14 [11 to 18]
  LT IgA GMFR - Day 14 | 4 [3 to 6] | 7 [5 to 9]
  LT IgA GMFR - Day 21 | 8 [5 to 11] | 12 [10 to 15]
  LT IgA GMFR - Day 28 | 12 [9 to 16] | 15 [12 to 18]
  LT IgA GMFR - Day 35 | 10 [7 to 15] | 13 [11 to 17]
  LT IgA GMFR - Day 194 | 5 [4 to 6] | 5 [4 to 7]

3. Primary Outcome: Seroconversion After a Self-administered LT Vaccine Patch (In-clinic or Away From Clinic) Compared to a Clinician-administered LT Vaccine Patch.
Description: The primary endpoint of this trial was to compare the immunogenicity (i.e., GMTs, GMFRs and seroconversion rates (SCR) for LT IgG and IgA) of subject self-administered [second] vaccination with clinician-administered [second] vaccination, using the deltoid/thigh (Vaccination 1/Vaccination 2) treatment regimen.
  seroconversion (SC): two-fold or greater rise in titer relative to Day 0 for LT IgG and a four-fold or greater rise in titer relative to Day 0 for LT IgA
Time Frame: Day 14, Day 21, Day 28, Day 35, Day 194
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of study participants
Arm/Group | Clinician Administered (Deltoid/ Thigh) | Self Administered (In-clinic & Non-clinic)
Number analyzed (Participants) | 41 | 80
percentage of study participants
  LT IgG SCR - Day 14 | 65 [48 to 79] | 73 [61 to 82]
  LT IgG SCR - Day 21 | 92 [79 to 98] | 98 [91 to 100]
  LT IgG SCR - Day 28 | 98 [87 to 100] | 99 [93 to 100]
  LT IgG SCR - Day 35 | 100 [91 to 100] | 99 [93 to 100]
  LT IgG SCR - Day 194 | 97 [87 to 100] | 100 [95 to 100]
  LT IgA SCR - Day 14 | 48 [32 to 64] | 59 [47 to 70]
  LT IgA SCR - Day 21 | 69 [52 to 83] | 85 [75 to 92]
  LT IgA SCR - Day 28 | 83 [67 to 93] | 90 [81 to 96]
  LT IgA SCR - Day 35 | 80 [64 to 91] | 87 [77 to 94]
  LT IgA SCR - Day 194 | 69 [52 to 83] | 62 [50 to 73]

4. Secondary Outcome: Number of Adverse Events for Self-administered LT Vaccine Patch and Comparison to the Clinician-administered LT Vaccine Patch
Time Frame: 6 months
Population: Number analyzed in the Outcome Measure Data Teble are the number of subjects with events
Measure: Number; unit: Events
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 40 | 40 | 40 | 40
Events
  All AEs | 347 | 358 | 358 | 387
  Local AEs: number analyzed (Participants) | 40 | 40 | 39 | 40
  Local AEs | 284 | 283 | 268 | 304
  Systemic AEs: number analyzed (Participants) | 21 | 26 | 29 | 30
  Systemic AEs | 63 | 75 | 90 | 83
  All Severe AEs: number analyzed (Participants) | 2 | 6 | 1 | 4
  All Severe AEs | 3 | 9 | 2 | 7
  Severe Local AEs: number analyzed (Participants) | 0 | 0 | 0 | 0
  Severe Systemic AEs: number analyzed (Participants) | 2 | 6 | 1 | 4
  Severe Systemic AEs | 3 | 9 | 2 | 7
  All Related AEs | 299 | 297 | 285 | 334
  Related Local AEs: number analyzed (Participants) | 40 | 40 | 39 | 40
  Related Local AEs | 284 | 283 | 268 | 304
  Related Systemic AEs: number analyzed (Participants) | 10 | 10 | 13 | 14
  Related Systemic AEs | 15 | 14 | 17 | 30
  All Serious AEs: number analyzed (Participants) | 1 | 3 | 0 | 0
  All Serious AEs | 2 | 3 |  |
  Serious Local AEs: number analyzed (Participants) | 0 | 0 | 0 | 0
  Serious Systemic AEs: number analyzed (Participants) | 1 | 3 | 0 | 0
  Serious Systemic AEs | 2 | 3 |  |

5. Secondary Outcome: Evaluation of Immunogenicity (GMT) for Deltoid/Thigh (Prime/Boost) Versus Deltoid/Deltoid Administered LT Vaccine.
Time Frame: 6 months
Population: The Overall Number of Participants Analyzed are the number of subjects in the ITT Population in each group. The number analyzed in the Outcome Measure Data Table are the number of subjects with non-missing data at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- Clinician-administered - Group 1: 1. st vaccination: administered by clinician; location: deltoid
  2. nd vaccination: administered by clinician; location: deltoid
- Clinician Administered (Deltoid/ Thigh) - Group 2: 1. st vaccination: administered by clinician; location: deltoid
  2. nd vaccination: administered by clinician; location: thigh
Arm/Group | Clinician-administered - Group 1 | Clinician Administered (Deltoid/ Thigh) - Group 2
Number analyzed (Participants) | 40 | 41
titers
  LT IgG Day 0 - GMT | 411 [302 to 561] | 362 [265 to 493]
  LT IgG Day 14 - GMT | 2176 [1326 to 3571] | 1974 [1203 to 3240]
  LT IgG Day 21 - GMT: number analyzed (Participants) | 40 | 39
  LT IgG Day 21 - GMT | 6292 [4136 to 9173] | 4747 [3241 to 6954]
  LT IgG Day 28 - GMT | 8895 [6453 to 12263] | 11153 [8090 to 15375]
  LT IgG Day 35 - GMT | 12460 [9639 to 16106] | 12165 [9410 to 15725]
  LT IgG Day 194 - GMT: number analyzed (Participants) | 40 | 39
  LT IgG Day 194 - GMT | 6694 [5095 to 8795] | 4997 [3790 to 6589]
  LT IgA Day 0 - GMT | 43 [33 to 56] | 54 [41 to 70]
  LT IgA Day 14 - GMT | 239 [155 to 368] | 218 [142 to 337]
  LT IgA Day 21 - GMT: number analyzed (Participants) | 40 | 39
  LT IgA Day 21 - GMT | 502 [358 to 703] | 430 [306 to 605]
  LT IgA Day 28 - GMT | 610 [444 to 839] | 632 [460 to 869]
  LT IgA Day 35 - GMT | 567 [419 to 767] | 548 [405 to 742]
  LT IgA Day 194 - GMT: number analyzed (Participants) | 40 | 39
  LT IgA Day 194 - GMT | 272 [206 to 360] | 254 [192 to 337]

6. Secondary Outcome: Safety for Self-administration In-clinic Compared to Self-administration Away From the Clinic.
Time Frame: 6 months
Population: Number Analyzed in Outcome Measure Data Table: in Group 3 only 39 subjects received the second vaccination.
Measure: Number; unit: Events
Arm/Group | Group 3 | Group 4
Number analyzed (Participants) | 40 | 40
Events
  Erythema - 1st vaccination | 37 | 38
  Erythema - 2nd vaccination: number analyzed (Participants) | 39 | 40
  Erythema - 2nd vaccination | 33 | 36
  Rash - 1st vaccination | 35 | 38
  Rash - 2nd vaccination: number analyzed (Participants) | 39 | 40
  Rash - 2nd vaccination | 20 | 23
  Pruritus - 1st vaccination | 37 | 31
  Pruiruts - 2nd vaccination: number analyzed (Participants) | 39 | 40
  Pruiruts - 2nd vaccination | 23 | 29
  Hyperpigmentation - 1st vaccination | 16 | 23
  Hyperpigmentation - 2nd vaccination: number analyzed (Participants) | 39 | 40
  Hyperpigmentation - 2nd vaccination | 7 | 14
  Edema - 1st vaccination | 5 | 5
  Edema - 2nd vaccination: number analyzed (Participants) | 39 | 40
  Edema - 2nd vaccination | 7 | 5
  Pain - 1st vaccination | 6 | 8
  Pain - 2nd vaccination: number analyzed (Participants) | 39 | 40
  Pain - 2nd vaccination | 5 | 4
  Fever - 1st vaccination | 1 | 0
  Fever - 2nd vaccination: number analyzed (Participants) | 39 | 40
  Fever - 2nd vaccination | 0 | 1
  Malaise - 1st vaccination | 3 | 4
  Malaise - 2nd vaccination: number analyzed (Participants) | 39 | 40
  Malaise - 2nd vaccination | 3 | 3
  Headache - 1st vaccination | 7 | 5
  Headache - 2nd vaccination: number analyzed (Participants) | 39 | 40
  Headache - 2nd vaccination | 9 | 4
  Diarrhea - 1st vaccination | 6 | 4
  Diarrhea - 2nd vaccination: number analyzed (Participants) | 39 | 40
  Diarrhea - 2nd vaccination | 3 | 4

7. Secondary Outcome: Evaluation of Immunogenicity (GMT) for Self-administration In-clinic Compared to Self-administration Away From the Clinic.
Time Frame: 6 months
Population: Overall Number of Participants Analyzed are the number of subjects in the ITT Population in each group. The Number analyzed in the Outcome Measure Data Table are the number of subjects with non-missing data at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 3 | Group 4
Number analyzed (Participants) | 40 | 40
titers
  LT IgG Day 0 - GMT | 473 [347 to 644] | 413 [303 to 564]
  LT IgG Day 14 - GMT | 2539 [1547 to 4166] | 3304 [2013 to 5422]
  LT IgG Day 21 - GMT: number analyzed (Participants) | 39 | 40
  LT IgG Day 21 - GMT | 6511 [4444 to 9537] | 8712 [5976 to 12701]
  LT IgG Day 28 - GMT: number analyzed (Participants) | 39 | 40
  LT IgG Day 28 - GMT | 10496 [7582 to 14528] | 14083 [10216 to 19414]
  LT IgG Day 35 - GMT: number analyzed (Participants) | 39 | 38
  LT IgG Day 35 - GMT | 11995 [9249 to 15556] | 13564 [10424 to 17651]
  LT IgG Day 194 - GMT: number analyzed (Participants) | 39 | 37
  LT IgG Day 194 - GMT | 5712 [4332 to 7532] | 6396 [4815 to 8495]
  LT IgA Day 0 - GMT | 54 [42 to 70] | 52 [40 to 68]
  LT IgA Day 21 - GMT: number analyzed (Participants) | 39 | 40
  LT IgA Day 21 - GMT | 549 [390 to 772] | 742 [530 to 1039]
  LT IgA Day 28 - GMT: number analyzed (Participants) | 39 | 40
  LT IgA Day 28 - GMT | 660 [478 to 911] | 891 [648 to 1225]
  LT IgA Day 35 - GMT: number analyzed (Participants) | 39 | 38
  LT IgA Day 35 - GMT | 605 [445 to 821] | 842 [618 to 1148]
  LT IgA Day 194 - GMT: number analyzed (Participants) | 39 | 37
  LT IgA Day 194 - GMT | 246 [186 to 327] | 338 [253 to 452]

8. Secondary Outcome: Evaluation of Immunogenicity (GMFR) for Deltoid/Thigh (Prime/Boost) Versus Deltoid/Deltoid Administered LT Vaccine
Time Frame: 6 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: fold change
Arm/Group | Clinician-administered - Group 1 | Clinician Administered (Deltoid/ Thigh) - Group 2
Number analyzed (Participants) | 40 | 41
fold change
  LT IgG Day 14 - GMFR | 5 [4 to 8] | 6 [4 to 8]
  LT IgG Day 21 - GMFR: number analyzed (Participants) | 40 | 39
  LT IgG Day 21 - GMFR | 15 [10 to 23] | 14 [9 to 20]
  LT IgG Day 28 - GMFR | 22 [15 to 32] | 31 [21 to 46]
  LT IgG Day 35 - GMFR | 30 [21 to 44] | 34 [23 to 49]
  LT IgG Day 194 - GMFR | 16 [12 to 23] | 14 [10 to 20]
  LT IgA Day 14 - GMFR | 6 [4 to 8] | 4 [3 to 6]
  LT IgA Day 21 - GMFR: number analyzed (Participants) | 40 | 39
  LT IgA Day 21 - GMFR | 12 [8 to 16] | 8 [5 to 11]
  LT IgA Day 28 - GMFR | 14 [10 to 19] | 12 [9 to 16]
  LT IgA Day 35 - GMFR | 13 [10 to 18] | 10 [8 to 14]
  LT IgA Day 194 - GMFR: number analyzed (Participants) | 40 | 39
  LT IgA Day 194 - GMFR | 6 [5 to 8] | 5 [4 to 6]

9. Secondary Outcome: Evaluation of Immunogenicity (SCR) for Deltoid/Thigh (Prime/Boost) Versus Deltoid/Deltoid Administered LT Vaccine
Time Frame: 6 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Clinician-administered - Group 1 | Clinician Administered (Deltoid/ Thigh) - Group 2
Number analyzed (Participants) | 40 | 41
Percent of Participants
  LT IgG Day 14 - SCR | 70 [54 to 83] | 65 [48 to 79]
  LT IgG Day 21 - SCR: number analyzed (Participants) | 40 | 39
  LT IgG Day 21 - SCR | 90 [76 to 97] | 92 [79 to 98]
  LT IgG Day 28 - SCR | 98 [87 to 100] | 97 [87 to 100]
  LT IgG Day 35 - SCR | 95 [83 to 99] | 100 [91 to 100]
  LT IgG Day 194 - SCR: number analyzed (Participants) | 40 | 39
  LT IgG Day 194 - SCR | 98 [87 to 100] | 97 [87 to 100]
  LT IgA Day 14 - SCR | 50 [34 to 66] | 48 [32 to 64]
  LT IgA Day 21 - SCR: number analyzed (Participants) | 40 | 39
  LT IgA Day 21 - SCR | 80 [64 to 91] | 69 [52 to 83]
  LT IgA Day 28 - SCR | 88 [73 to 96] | 83 [67 to 93]
  LT IgA Day 35 - SCR | 90 [76 to 97] | 80 [64 to 91]
  LT IgA Day 194 - SCR: number analyzed (Participants) | 40 | 39
  LT IgA Day 194 - SCR | 70 [54 to 83] | 69 [52 to 83]

10. Secondary Outcome: Evaluation of Immunogenicity (GMFR) for Self-administration In-clinic Compared to Self-administration Away From the Clinic
Time Frame: 6 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: fold change
Arm/Group | Group 3 | Group 4
Number analyzed (Participants) | 40 | 40
fold change
  Lt IgG Day 14 - GMFR | 5 [4 to 8] | 8 [5 to 12]
  LT IgG Day 21 - GMFR: number analyzed (Participants) | 39 | 40
  LT IgG Day 21 - GMFR | 14 [9 to 21] | 21 [14 to 31]
  LT IgG Day 28 - GMFR: number analyzed (Participants) | 39 | 40
  LT IgG Day 28 - GMFR | 22 [15 to 33] | 34 [23 to 50]
  LT IgG Day 35 - GMFR: number analyzed (Participants) | 39 | 38
  LT IgG Day 35 - GMFR | 26 [18 to 37] | 34 [23 to 49]
  LT IgG Day 194 - GMFR: number analyzed (Participants) | 39 | 37
  LT IgG Day 194 - GMFR | 12 [9 to 17] | 16 [11 to 23]
  LT IgA Day 14 - GMFR | 6 [4 to 9] | 8 [5 to 12]
  LT IgA Day 21 - GMFR: number analyzed (Participants) | 39 | 40
  LT IgA Day 21 - GMFR | 10 [7 to 14] | 14 [10 to 20]
  LT IgA Day 28 - GMFR: number analyzed (Participants) | 39 | 40
  LT IgA Day 28 - GMFR | 12 [9 to 17] | 17 [13 to 23]
  LT IgA Day 35 - GMFR: number analyzed (Participants) | 39 | 38
  LT IgA Day 35 - GMFR | 11 [8 to 15] | 16 [12 to 22]
  LT IgA Day 194 - GMFR: number analyzed (Participants) | 39 | 37
  LT IgA Day 194 - GMFR | 5 [4 to 6] | 6 [5 to 8]

11. Secondary Outcome: Evaluation of Immunogenicity (SCR) for Self-administration In-clinic Compared to Self-administration Away From the Clinic
Time Frame: 6 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Group 3 | Group 4
Number analyzed (Participants) | 40 | 40
Percent of Participants
  LT IgG Day 14 - SCR | 68 [51 to 81] | 78 [62 to 90]
  LT IgG Day 21 - SCR: number analyzed (Participants) | 39 | 40
  LT IgG Day 21 - SCR | 97 [87 to 100] | 98 [87 to 100]
  LT IgG Day 28 - SCR: number analyzed (Participants) | 39 | 40
  LT IgG Day 28 - SCR | 100 [91 to 100] | 98 [87 to 100]
  LT IgG Day 35 - SCR: number analyzed (Participants) | 39 | 38
  LT IgG Day 35 - SCR | 100 [91 to 100] | 97 [86 to 100]
  LT IgG Day 194 - SCR: number analyzed (Participants) | 39 | 37
  LT IgG Day 194 - SCR | 100 [91 to 100] | 100 [91 to 100]
  LT IgA Day 14 - SCR | 58 [41 to 73] | 60 [43 to 75]
  LT IgA Day 21 - SCR: number analyzed (Participants) | 39 | 40
  LT IgA Day 21 - SCR | 84 [70 to 94] | 85 [70 to 94]
  LT IgA Day 28 - SCR: number analyzed (Participants) | 39 | 40
  LT IgA Day 28 - SCR | 92 [79 to 98] | 88 [73 to 96]
  LT IgA Day 35 - SCR: number analyzed (Participants) | 39 | 38
  LT IgA Day 35 - SCR | 85 [70 to 94] | 90 [75 to 97]
  LT IgA Day 194 - SCR: number analyzed (Participants) | 39 | 37
  LT IgA Day 194 - SCR | 56 [40 to 72] | 68 [50 to 82]

ADVERSE EVENTS:
Arm/Group | Clinician Administered (Deltoid) | Clinician Administered (Thigh) | Self Administered (In-clinic) | Self Administered (Non-clinic)
Serious Adverse Events (participants affected / at risk) | 1/40 | 3/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 40/40 | 40/40 | 40/40 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinician Administered (Deltoid) (N=40) | Clinician Administered (Thigh) (N=40) | Self Administered (In-clinic) (N=40) | Self Administered (Non-clinic) (N=40)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brugada syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clinician Administered (Deltoid) (N=40) | Clinician Administered (Thigh) (N=40) | Self Administered (In-clinic) (N=40) | Self Administered (Non-clinic) (N=40)
Diarrhea (Gastrointestinal disorders) | 2 | 8 | 7 | 6
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Malaise (General disorders) | 3 | 3 | 6 | 7
Influenza (Infections and infestations) | 1 | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 5 | 2 | 4 | 5
Sinusitis (Infections and infestations) | 0 | 2 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 5 | 2
Application site discoloration (Injury, poisoning and procedural complications) | 26 | 30 | 20 | 29
Application site erythema (Injury, poisoning and procedural complications) | 39 | 38 | 37 | 39
Application site edema (Injury, poisoning and procedural complications) | 9 | 12 | 11 | 8
Application site excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 0
Application site pain (Injury, poisoning and procedural complications) | 12 | 8 | 10 | 9
Application site pruritus (Injury, poisoning and procedural complications) | 39 | 36 | 37 | 35
Application site rash (Injury, poisoning and procedural complications) | 38 | 38 | 35 | 38
Application site scab (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 4
Blood glucose increased (Investigations) | 0 | 3 | 2 | 3
Protein urine present (Investigations) | 2 | 1 | 1 | 0
Red blood cells in urine (Investigations) | 8 | 3 | 7 | 4
Headache (Nervous system disorders) | 6 | 9 | 12 | 8
Hematuria (Renal and urinary disorders) | 1 | 0 | 2 | 1
Proteinuria (Renal and urinary disorders) | 1 | 2 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other